CLINICAL TRIAL: NCT03560297
Title: SeRenade Parent-Child Music Class Program for Families of Children With and Without ASD
Brief Title: SeRenade Parent-Child Music Class Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Endowment for the Arts, United States (U.S. Federal Agency)
Responsible Party: Principal Investigator, Miriam Lense, Research Instructor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 160784
Record Dates: First submitted 2018-05-21; First posted 2018-06-18 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SeRenade Program (Experimental): Parent-Child Music Class Program (parent training, peer inclusion, musical play)
  Interventions: Behavioral: SeRenade Parent-Child Music Class
- Delayed/Waitlist Program (Experimental): Participants do not participate in the program for a time period
  Interventions: Behavioral: Delayed Intervention

INTERVENTIONS:
Behavioral: SeRenade Parent-Child Music Class — Parent-Child Music Class involving parent training, peer inclusion, and musical play
  Arms: SeRenade Program
Behavioral: Delayed Intervention — Participants receive intervention after delay
  Arms: Delayed/Waitlist Program

SUMMARY:
This pilot study examines the impact of the SeRenade Parent-Child Music Class Program, which emphasizes parent training, peer inclusion, and musical play combined with established behavioral techniques, on the development of child social engagement, positive behavior, and parental well-being.

DETAILED DESCRIPTION:
This pilot study evaluates the impact of the SeRenade Parent-Child Music Class Program on families of children with and without autism spectrum disorders (ASD). This study examines the impact of this program on social development in children with ASD, parental stress and efficacy, and parent-child relationships. A primary goal of this study is to examine multiple levels of analysis including families' experience within and outside of the music class program.

ELIGIBILITY:
Inclusion Criteria:

* children diagnosed with ASD or children without ASD

Exclusion Criteria:

* currently enrolled in music therapy or parent-child music classes (for children with ASD); significant behavior problems (e.g., aggression toward other children); significant hearing or visual impairments

Ages: 20 Months to 72 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2020-03-20 (Actual)

PRIMARY OUTCOMES:
Motor Imitation Scale | Change from pre to post program (baseline and 12-weeks)
  Standardized elicited imitation assessment; scores range 0-32; greater scores indicate greater imitation skills
Actions & Gestures | Change from pre to post program (baseline and 12-weeks)
  Standardized parent report questionnaire of child's gestures/actions/pretend play
Parenting Stress Index, 4th edition Short Form | Change from pre to post program (baseline and 12-weeks)
  Standardized parent report questionnaire
Parenting Efficacy/Quality | Change from pre to post program (baseline and 12-weeks)
  Parent report questionnaire; higher scores indicate greater efficacy, range 10-40

SECONDARY OUTCOMES:
Parent-Child Interaction | Change from pre to post program (baseline and 12-weeks)
  parent-child play/music session
social visual attention eye-tracking paradigm | Change from pre to post program (baseline and 12-weeks)

OTHER OUTCOMES:
parent mood/connection | change from before/after the class session at class 1 (week 1) to 12 (week 12) (a session of classes is 12-weeks on average)
  parent ratings
Program acceptability | post program (12 weeks)
  parent program evaluation survey

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided
Deidentified data and codebooks will be available to researchers upon request.

REFERENCES:
- [Derived] Geretsegger M, Fusar-Poli L, Elefant C, Mossler KA, Vitale G, Gold C. Music therapy for autistic people. Cochrane Database Syst Rev. 2022 May 9;5(5):CD004381. doi: 10.1002/14651858.CD004381.pub4. PMID 35532041